CLINICAL TRIAL: NCT06523933
Title: Distribution of Bacteria in Otitis Media With Effusion After Radiotherapy For Nasopharyngeal Carcinoma.
Brief Title: Distribution of Bacteria in OME After Radiotherapy For NPC.
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-448-01
Record Dates: First submitted 2024-07-10; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media Effusion; Nasopharyngeal Carcinoma
Keywords: Otitis Media Effusion; Nasopharyngeal Carcinoma; Bacteria
MeSH Terms: conditions — Otitis Media with Effusion; Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — middle ear effusion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- ON+: Patients with OME after NPC with a Positive Result of Bacteria Culture of Middle Ear Effusion.
- ON-: Patients with OME after NPC with a Negative Result of Bacteria Culture of Middle Ear Effusion.
- O+: Patients with OME with a Positive Result of Bacteria Culture of Middle Ear Effusion.
- O-: Patients with OME with a Negative Result of Bacteria Culture of Middle Ear Effusion.

SUMMARY:
To observe the prognostic difference of tympanocentesis in different kinds of otitis media effusion.

DETAILED DESCRIPTION:
This study is a prospective, observational clinical study to observe the difference in prognosis of tympanocentesis in different kinds of otitis media effusion (OME), especially OME after radiotherapy for nasopharyngeal carcinoma (NPC). A total of 234 patients diagnosed with OME who are given the treatment of tympanocentesis only, including outpatient and inpatient patients, were included in the study. The middle ear effusion collected during the tympanocentesis is sent for bacterial culture. The positive rate of the effusion and the recurrence rate within 24 weeks will be compared in order to figure out whether bacterial infection is an important influencing factor for some kinds of OME in addition to eustachian tube dysfunction, which is acknowledged.

ELIGIBILITY:
Inclusion Criteria:

* patients clinical diagnosis of OME or OME after radiotherapy for NPC (Diagnostic criteria: fluid visible in the middle ear and a type B tympanogram).
* patients volunteered to participate in the study and signed the informed consent

Exclusion Criteria:

* NPC recurrence or other malignant tumor after radiotherapy.
* clear diagnosis of Eustachian ostium atresia or nasal obstruction diseases, such as severe deviated nasal septum, choanal atresia, osteoradionecrosis of skull base after radiotherapy, etc.
* pregnant and lactating women.
* patients with severe underlying diseases or with severe liver and kidney dysfunction.
* patients who could not cooperate (including poor hearing and radiation encephalopathy)
* patients with other middle ear diseases, such as middle ear cholesteatoma, osteoradionecrosis of temporal bone after radiotherapy, etc.
* severe deglutition disorders
* cleft palate

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with OME and OME after radiotherapy for NPC, who are given the treatment of tympanostomy only, including outpatient and inpatient patients, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-11-12 (Estimated); Study Completion 2025-05-12 (Estimated)

PRIMARY OUTCOMES:
Positive Bacterial Culture Rate in Middle Ear Effusion | Up to 24 weeks

SECONDARY OUTCOMES:
Changes in Air Pressure (Tympanogram) | Collected at 6, 12, 24 Weeks after Tympanocentesis
  Tympanogram changed from type B to type A or type C.
Eustachian Tube Dysfunction Questionnaire (ETDQ-7) | Collected at 6, 12, 24 Weeks after Tympanocentesis
  The ETDQ-7 tool is used to assess the symptoms of Otitis Media With Effusion (OME), which consists of seven items with a scale of graduated responses ranging from 1 (No Problem) to 7 (Severe Problem), and 4 would correspond to a Moderate Problem. If the total score is more than 14, it is considered that there is eustachian tube dysfunction. The average post-operative ETDQ-7 score is less than 2.1 or decrease > 0.5 (minimal clinically important difference=0.5), it is considered that the eustachian tube function is improved.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Xiong, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China